CLINICAL TRIAL: NCT01342952
Title: An Open-label, Long Term Extension Study for Treatment of Pulmonary Arterial Hypertension in Paediatric Patients Aged 8 Years up to 18 Years Who Have Participated in AMB112529 and in Whom Continued Treatment With Ambrisentan is Desired
Brief Title: Long-term Ambrisentan Extension Study for Pediatric Patients Who Participated in AMB112529
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114588; 2010-021572-29 (EudraCT Number)
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Results first posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Hypertension, Pulmonary
Keywords: pulmonary arterial hypertension; pediatrics
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — ambrisentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ambrisentan (Experimental): Open label, flexible dosing from 2.5 mg to 10 mg (not to exceed 0.25 mg/kg) per day
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan — open label, flexible dosing from 2.5 to 10 mg (not to exceed 10 mg/kg) per day

SUMMARY:
An open label, long term extension to Study AMB112529. All subjects may remain in the extension study for a minimum of six months. Beyond the six month period, subjects may continue in the extension study until one of the following conditions is met:

the subject turns 18 years of age (when the subject can receive marketed product) the product is approved and available for use in the subject's age group, development for use in the paediatric population is discontinued. the subject decides he/she no longer wants to participate in the study, the investigator considers it is in the best interest of the subject to discontinue ambrisentan (e.g. for safety reasons).

The primary objective is the long-term safety and tolerability of ambrisentan in the paediatric PAH population. Secondary objectives are all cause mortality and change from baseline in Study AMB112529 on efficacy parameters.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a rare, progressive, highly debilitating disease characterized by vascular obstruction and the variable presence of vasoconstriction, leading to increased pulmonary vascular resistance and right-sided heart failure. If left untreated, PAH ultimately leads to right ventricular failure and death; adult subjects have a median survival of 2.8 years without treatment. Epidemiological estimates vary but prevalence in Europe is thought to be of the order of 15 cases per million. Large scale epidemiology studies of PAH in children have not been conducted and there is no or limited outcome data in paediatric PAH patients. A register in France (1995-1996) estimates the prevalence in children is as low as 3.7 cases per million. In a national, comprehensive country wide survey of the epidemiology of idiopathic PAH (IPAH) management and survival in the United Kingdom (UK) the incidence was 0.48 cases per million children per year and the prevalence was 2.1 cases per million children.

Ambrisentan (VOLIBRIS™ tablets) is an endothelin receptor antagonist (ERA) marketed in the European Union (EU) and some other countries by GlaxoSmithKline (GSK) and in the United States as LETAIRIS® by Gilead Sciences Inc. Ambrisentan is indicated for the treatment of adult patients with PAH to improve exercise capacity, decrease the symptoms of PAH, and delay clinical worsening.

The primary purpose of this long term paediatric study is to provide clinically relevant information on the long term safety of ambrisentan in children with the most common causes of PAH in this age group. This study is only open to patients who have participated in Study AMB112529, A randomized, open label study comparing safety and efficacy parameters for a high and a low dose of ambrisentan (adjusted for body weight) for the treatment of pulmonary arterial hypertension in paediatric patients aged 8 years up to 18 years, and in whom continued treatment with ambrisentan is warranted.

This study is part of a Paediatric Investigational Plan (PIP; EMEA-000434-PIP01-08) agreed with the European Medicines Agency's Paediatric Committee (PDCO).

ELIGIBILITY:
Inclusion Criteria:

* Have participated in and complied, to the best of their ability, with the protocol for AMB112529 and have met one of the following:

  1. Completed the Week 24 visit in AMB112529;
  2. Required additional targeted treatment for PAH due to inadequate response to the current treatment or worsening of their clinical condition prior to week 24 in AMB112529;
  3. Required reduction in dose of baseline targeted treatment for PAH after ambrisentan was added to the treatment regimen;
  4. In the opinion of the investigator, continued treatment with ambrisentan is warranted.
* A female is eligible to participate in this study, as assessed by the investigator, if she is of:

  1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or,
  2. Child-bearing potential - has a negative pregnancy test and is not lactating and, if sexually active, agrees to continue to use 2 reliable methods of contraception until study completion and for at least 30 days following the last dose of study drug (reliable methods of contraception are listed in Appendix 2).
* Subject or subject's legal guardian is able and willing to give written informed consent. As part of the consent, female subjects of childbearing potential will be informed of the risk of teratogenicity and will need to be counselled in a developmentally appropriate manner on the importance of pregnancy prevention; and male subjects will need to be informed of potential risk of testicular tubular atrophy and aspermia.

Exclusion Criteria:

* Subjects who were withdrawn from ambrisentan in Study AMB112529;
* Subjects who did not comply with the protocol in Study AMB112529;
* Female subjects who are pregnant or breastfeeding;
* Subjects with severe renal impairment (estimated creatinine clearance <30 mL/min assessed within the previous 45 days) at the point of transition from Study AMB112529 into this study;
* Subject with clinically significant fluid retention in the opinion of the investigator;
* Subject with clinically significant anaemia in the opinion of the investigator;
* Subjects who are to enter another clinical trial or be treated with another investigational product after exiting Study AMB112529.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2011-06-21 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- United States (4):
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, New York, New York
- Argentina (3):
  - GSK Investigational Site, Guymallen, Mendoza Province
  - GSK Investigational Site, Ciudad de Buenos Aires
  - GSK Investigational Site, Córdoba
- France (3):
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Toulouse
- Germany (2):
  - GSK Investigational Site, Giessen, Hesse
  - GSK Investigational Site, Berlin
- GSK Investigational Site, Budapest, Hungary
- Italy (2):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, San Donato Milanese (MI), Lombardy
- Japan (2):
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Russia (3):
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
- GSK Investigational Site, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label, long term extension of study AMB112529 (NCT01342952) which evaluated safety and tolerability of ambrisentan in the pediatric (aged 8 years up to 18 years) Pulmonary Arterial Hypertension (PAH) population.
Pre-assignment Details: A total of 38 participants were enrolled in this study.
Groups:
- Ambrisentan 2.5 mg (ITT): Participants received ambrisentan 2.5 milligrams (mg) dose of ambrisentan orally in tablet/s form once daily. The Intent-to-Treat (ITT) Population consisted of all participants who received at least 1 dose of study drug. Participants were considered as belonging to ITT treatment group at the start of study AMB114588.
- Ambrisentan 5 mg (ITT): Participants received 5 mg dose of ambrisenten orally in tablet form once daily. The ITT Population consisted of all participants who received at least 1 dose of study drug. Participants were considered as belonging to ITT treatment group at the start of study AMB114588.
- Ambrisentan 7.5 mg (ITT): Participants received 7.5 mg dose of ambrisentan orally in tablet/s form once daily. The ITT Population consisted of all participants who received at least 1 dose of study drug. Participants were considered as belonging to ITT treatment group at the start of study AMB114588.
- Ambrisentan 10 mg (ITT): Participants received 10 mg dose of ambrisentan orally in tablet/s form once daily. The ITT Population consisted of all participants who received at least 1 dose of study drug. Participants were considered as belonging to ITT treatment group at the start of study AMB114588.
Period: Overall Study
Arm/Group | Ambrisentan 2.5 mg (ITT) | Ambrisentan 5 mg (ITT) | Ambrisentan 7.5 mg (ITT) | Ambrisentan 10 mg (ITT)
Started | 9 | 19 | 5 | 5
Intent-to-Treat Population (The Intention-to-Treat (ITT) Population consisted of all participants who received at least 1 dose of study drug. Participants were considered as belonging to ITT population at the start of study AMB114588) | 9 | 19 | 5 | 5
Safety Population (The Safety Population is defined as all participants who received at least 1 dose of study drug. Participants were considered as belonging to the treatment group according to the highest dose received) | 4 | 16 | 6 | 12
Completed | 5 | 8 | 3 | 5
Not Completed | 4 | 11 | 2 | 0
Not completed — Adverse Event | 0 | 5 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Physician Decision | 3 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were presented for ITT Population, consisted of all participants who received at least 1 dose of study drug. Participants were considered as belonging to ITT population at the start of study AMB114588
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambrisentan 2.5 mg (ITT) | Ambrisentan 5 mg (ITT) | Ambrisentan 7.5 mg (ITT) | Ambrisentan 10 mg (ITT) | Total
Number analyzed (Participants) | 9 | 19 | 5 | 5 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.7 (2.29) | 11.9 (2.57) | 12.6 (2.61) | 15.2 (0.84) | 11.9 (2.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 4 | 5 | 25
  Male | 2 | 10 | 1 | 0 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 1 | 1 | 0 | 0 | 2
  American Indian or Alaskan Native | 1 | 0 | 0 | 0 | 1
  Asian - Central/South Asian Heritage | 0 | 1 | 0 | 0 | 1
  Asian - East Asian Heritage | 0 | 1 | 0 | 0 | 1
  Asian - Japanese Heritage | 3 | 2 | 0 | 0 | 5
  Asian - South East Asian Heritage | 0 | 0 | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 4 | 14 | 4 | 5 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Treatment-emergent Adverse Events (Non-STEAEs) and Serious Treatment-emergent Adverse Events (STEAEs)
Description: AE was defined as any untoward medical occurrence in participant or clinical investigation participant,temporally associated with use of medicinal product, whether or not considered related to medicinal product.SAE was defined as any untoward medical occurrence that, at any dose: results in death,is life threatening, requires hospitalization or prolongation of existing hospitalization,results in disability or incapacity,or is congenital anomaly or birth defect, important medical events that may not immediately life threatening or result in death or hospitalization but may jeopardize participant or may require medical or surgical intervention as per medical or scientific judgement or associated with drug-induced liver injury.TEAE is any event that was not present prior to initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment. TEAEs which were not serious TEAEs were considered as non serious TEAEs.
Time Frame: Up to 10 years and 11 months
Population: Safety Population consisted of all participants who received at least 1 dose of study drug. Participants were considered as belonging to the treatment group according to the highest dose received in the extension study (AMB114588)
Measure: Count of Participants; unit: Participants
Groups:
- Ambrisentan 2.5 mg (Safety): Participants received ambrisentan 2.5 mg tablet orally once daily. The Safety Population consisted of all participants who received at least 1 dose of study drug. Participants were considered as belonging to the treatment group according to the highest dose received in the extension study (AMB114588).
- Ambrisentan 5 mg (Safety): Participants received ambrisentan 5 mg tablet orally once daily. The Safety Population consisted of all participants who received at least 1 dose of study drug. Participants were considered as belonging to the treatment group according to the highest dose received in the extension study (AMB114588).
- Ambrisentan 7.5 mg (Safety): Participants received ambrisentan 7.5 mg tablet orally once daily. The Safety Population consisted of all participants who received at least 1 dose of study drug. Participants were considered as belonging to the treatment group according to the highest dose received in the extension study (AMB114588).
- Ambrisentan 10 mg (Safety): Participants received ambrisentan 10 mg tablet orally once daily. The Safety Population consisted of all participants who received at least 1 dose of study drug. Participants were considered as belonging to the treatment group according to the highest dose received in the extension study (AMB114588).
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 16 | 6 | 12
Participants
  Non-STEAEs | 3 | 13 | 5 | 10
  STEAEs | 2 | 7 | 4 | 8

2. Primary Outcome: Change From Baseline in Liver Function Parameters: Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Gamma Glutamyl Transferase (GGT), Total Bilirubin
Description: Blood samples were collected from participants for analysis of following clinical chemistry parameters: ALT, AST, GGT, total bilirubin. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 10 | 5 | 9
Millimoles per liter
  ALT | -7.5 (12.56) | -1.0 (8.64) | 0.8 (4.09) | 4.0 (7.42)
  AST | -11.8 (6.29) | -5.6 (7.23) | -1.0 (2.55) | -2.1 (8.13)
  GGT | -0.5 (15.00) | -7.0 (10.45) | -0.8 (8.44) | -4.6 (28.30)
  Total bilirubin | -5.3 (12.47) | -4.0 (3.30) | -2.8 (6.06) | 3.1 (8.45)

3. Primary Outcome: Change From Baseline in Chemistry Parameters: Calcium, Chloride, Carbon Dioxide (CO2) Content, Glucose, Potassium, Magnesium, Sodium, Phosphorus Inorganic, Blood Urea Nitrogen (BUN)
Description: Blood samples were collected from participants for analysis of following clinical chemistry parameters: Calcium, chloride, CO2 content, glucose, potassium, magnesium, sodium, phosphorus inorganic, and BUN. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 3 | 10 | 5 | 9
Millimoles per liter
  Calcium | -0.150 (0.1769) | -0.054 (0.0779) | 0.028 (0.0630) | -0.060 (0.1075)
  Chloride | 1.7 (5.13) | 2.6 (1.65) | 0.4 (3.44) | -0.6 (2.96)
  CO2 content | -0.3 (2.89) | 2.2 (1.87) | 0.2 (3.70) | 0.0 (1.80)
  Glucose | 0.167 (0.4163) | -0.150 (1.1414) | 0.120 (0.5541) | 0.478 (0.9107)
  Potassium | -0.30 (0.529) | -0.07 (0.337) | -0.02 (0.148) | -0.12 (0.327)
  Magnesium | -0.100 (0.0872) | -0.062 (0.0898) | 0.028 (0.0683) | 0.012 (0.0716)
  Sodium | 2.7 (1.15) | 1.0 (1.63) | -0.2 (0.84) | 0.7 (1.87)
  Phosphorus inorganic | -0.340 (0.1311) | -0.159 (0.3055) | -0.212 (0.3440) | -0.108 (0.2408)
  BUN | -0.10 (1.808) | -0.51 (1.649) | -0.14 (1.274) | 0.33 (1.507)

4. Primary Outcome: Change From Baseline in Chemistry Parameters: Alkaline Phosphatase (ALP), Creatine Kinase (CK), Lactate Dehydrogenase (LDH)
Description: Blood samples were collected from participants for analysis of following clinical chemistry parameters: ALP, CK, LDH. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 3 | 10 | 5 | 9
International units per Liter
  ALP | -77.7 (57.01) | -109.5 (71.51) | -148.8 (151.78) | -135.6 (97.33)
  CK | -18.7 (23.07) | 4.0 (100.83) | 46.6 (89.55) | -9.7 (13.96)
  LDH | -40.3 (45.54) | -48.9 (71.64) | -12.8 (22.58) | -28.3 (37.23)

5. Primary Outcome: Change From Baseline in Chemistry Parameters: Creatinine, Uric Acid
Description: Blood samples were collected from participants for analysis of following clinical chemistry parameters: Creatinine, uric acid. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 3 | 10 | 5 | 9
Micromoles per liter
  Creatinine | 6.27 (19.775) | 8.16 (9.602) | 10.26 (8.008) | 19.31 (14.698)
  Uric acid | -64.67 (119.169) | -83.60 (90.103) | -45.40 (77.584) | 21.22 (79.330)

6. Primary Outcome: Change From Baseline in Chemistry Parameters: Albumin, Total Protein
Description: Blood samples were collected from participants for analysis of following clinical chemistry parameters: Albumin, total protein. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 3 | 10 | 5 | 9
Grams per liter
  Albumin | -3.3 (4.04) | -1.2 (3.16) | 1.6 (1.14) | -2.0 (4.42)
  Total protein | -3.7 (4.51) | -3.4 (4.93) | 3.0 (5.24) | -3.0 (7.33)

7. Primary Outcome: Change From Baseline in Hematology Parameters: Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC)
Description: Blood samples were collected from participants for analysis of following hematology parameters: Hemoglobin and MCHC. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per Liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 3 | 9 | 5 | 9
Grams per Liter
  Hemoglobin | -23.0 (38.63) | -4.7 (16.15) | 0.8 (9.71) | 1.3 (20.12)
  MCHC | -9.3 (16.01) | -12.4 (17.31) | -6.0 (12.98) | -1.1 (11.72)

8. Primary Outcome: Change From Baseline in Hematology Parameters: Hematocrit
Description: Blood samples were collected from participants for analysis of following hematology parameters: Hematocrit. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 3 | 9 | 5 | 9
Proportion of red blood cells in blood | -0.0610 (0.10235) | -0.0004 (0.04543) | 0.0100 (0.02884) | 0.0040 (0.06572)

9. Primary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils, White Blood Cells (WBC), Platelet Count
Description: Blood samples were collected from participants for analysis of following hematology parameters: Basophils, eosinophils, lymphocytes, monocytes, total neutrophils, WBC, platelet count. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per Liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 3 | 9 | 5 | 9
Giga cells per Liter
  Basophils | -0.007 (0.0153) | 0.019 (0.0417) | -0.006 (0.0152) | -0.002 (0.0148)
  Eosinophils | -0.210 (0.4139) | 0.034 (0.1096) | -0.026 (0.0602) | 0.009 (0.0746)
  Lymphocytes | -1.107 (0.7310) | -0.329 (1.1373) | -0.152 (0.6937) | -0.394 (1.1063)
  Monocytes | -0.013 (0.1550) | 0.040 (0.1273) | -0.006 (0.1635) | 0.037 (0.1986)
  Total neutrophils | 0.677 (1.9014) | -0.974 (1.2239) | 0.412 (0.6278) | 0.524 (2.0030)
  WBC | -0.67 (2.616) | -1.22 (2.072) | 0.22 (0.421) | 0.18 (2.787)
  Platelet count: number analyzed (Participants) | 3 | 9 | 5 | 7
  Platelet count | -34.0 (27.18) | -29.3 (50.03) | -9.2 (30.87) | -0.4 (64.78)

10. Primary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscle Hemoglobin
Description: Blood samples were collected from participants for analysis of following hematology parameter: Mean Corpuscle Hemoglobin. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 3 | 9 | 5 | 9
Picograms | -1.70 (3.315) | -1.46 (2.823) | -0.70 (1.512) | 0.11 (1.981)

11. Primary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscle Volume
Description: Blood samples were collected from participants for analysis of following hematology parameter: Mean Corpuscle Volume. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 3 | 9 | 5 | 9
Femtoliters | -2.3 (6.66) | -1.0 (5.52) | -0.8 (2.68) | 0.8 (5.61)

12. Primary Outcome: Change From Baseline in Hematology Parameters: Red Blood Cell Count, Reticulocytes
Description: Blood samples were collected from participants for analysis of following hematology parameters: Red Blood Cell count, reticulocytes. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 3 | 9 | 5 | 9
Trillion cells per liter
  Red Blood Cell count | -0.57 (0.862) | 0.07 (0.387) | 0.14 (0.251) | 0.00 (0.497)
  Reticulocytes | 0.01427 (0.024625) | -0.00816 (0.043615) | 0.00906 (0.013265) | 0.01843 (0.041832)

13. Primary Outcome: Number of Participants With Abnormal Values for Physical Examination Parameter: Liver Size
Description: Physical examination included measurement of liver size. Any abnormal enlargement or reduction in the size of the liver is reported. Liver size was assessed as normal or abnormal. Data for abnormal (improved, worsened and unchanged) liver size is presented. End of study visit data is presented.
Time Frame: Up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 10 | 5 | 10
Participants
  Liver Size: Abnormal: Improved | 0 | 0 | 0 | 0
  Liver Size: Abnormal: Worsened | 0 | 0 | 0 | 0
  Liver Size: Abnormal: Unchanged | 0 | 0 | 0 | 2

14. Primary Outcome: Number of Participants With Abnormal Values for Physical Examination Parameter: Jugular Venous Pressure
Description: Physical examination included measurement of Jugular venous pressure. Jugular venous pressure was assessed as normal or abnormal. Data for abnormal (improved, worsened and unchanged) jugular venous pressure is presented. End of study visit data is presented.
Time Frame: Up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 10 | 5 | 10
Participants
  Jugular Venous Pressure: Abnormal: Improved | 0 | 0 | 0 | 0
  Jugular Venous Pressure: Abnormal: Worsened | 0 | 0 | 0 | 0
  Jugular Venous Pressure: Abnormal: Unchanged | 0 | 0 | 0 | 2

15. Primary Outcome: Number of Participants With Abnormal Values for Physical Examination Parameters: Ascites
Description: Physical examination included measurement of ascites. Ascites were assessed as present or absent. Data for ascites present with improved, worsened and unchanged is presented. End of study visit data is presented.
Time Frame: Up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 10 | 5 | 10
Participants
  Ascites: Present: Improved | 0 | 0 | 0 | 0
  Ascites: Present: Worsened | 0 | 0 | 0 | 0
  Ascites: Present: Unchanged | 0 | 0 | 0 | 2

16. Primary Outcome: Number of Participants With Abnormal Values for Physical Examination Parameter: Peripheral Edema
Description: Physical examination included measurement of peripheral edema. Peripheral edema were assessed as present or absent. Data for peripheral edema present with improved, worsened and unchanged is presented. End of study visit data is presented.
Time Frame: Up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 10 | 5 | 10
Participants
  Peripheral edema: Present: Improved | 0 | 0 | 0 | 0
  Peripheral edema: Present: Worsened | 0 | 0 | 0 | 0
  Peripheral edema: Present: Unchanged | 0 | 0 | 0 | 0

17. Primary Outcome: Percentage of Saturated Oxygen Level (Physical Examination Parameter)
Description: Physical examination included measurement of saturated oxygen. End of study visit data is presented.
Time Frame: Up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 10 | 5 | 10
Percentage of oxygen saturation | 95.5 (4.20) | 96.8 (2.04) | 97.4 (1.34) | 96.9 (1.97)

18. Primary Outcome: Change From Baseline in Vital Signs Parameter: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP was measured for the participants at indicated time points. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 10 | 5 | 10
Millimeters of mercury
  SBP | 16.3 (16.38) | 8.4 (17.99) | 1.2 (18.63) | 8.5 (12.22)
  DBP | 1.5 (5.80) | 2.3 (12.70) | 3.6 (16.96) | 2.1 (9.67)

19. Primary Outcome: Change From Baseline in Vital Signs Parameter: Heart Rate
Description: Heart rate was measured for the participants at indicated time points. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 10 | 5 | 10
Beats per minute | -9.0 (13.44) | -4.0 (8.08) | -3.8 (11.50) | -6.0 (15.06)

20. Primary Outcome: Change From Baseline in Vital Signs Parameter: Weight
Description: Weight was measured for the participants at indicated time points. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 10 | 5 | 10
Kilograms | 17.43 (12.695) | 10.73 (8.628) | 7.12 (5.346) | 12.17 (16.300)

21. Primary Outcome: Change From Baseline in Vital Sign Parameter: Height
Description: Height was measured for the participants at indicated time points. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 10 | 5 | 10
Centimeters | 25.3 (19.99) | 9.9 (9.92) | 7.2 (9.47) | 12.1 (17.55)

22. Primary Outcome: Change From Baseline in Vital Sign Parameter: Body Mass Index
Description: Body mass index was measured for the participants at indicated time points. Body mass index was calculated as weight in kilograms (kg) divided by the square of their height in meters (m^2). Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Kilogram per meter square
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 10 | 5 | 10
Kilogram per meter square | 2.65 (2.195) | 2.45 (1.828) | 1.52 (1.633) | 1.99 (2.642)

23. Primary Outcome: Change From Baseline in Vital Sign Parameter: Body Surface Area
Description: Body surface area was measured for the participants at indicated time points. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Meter square
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 10 | 5 | 10
Meter square | 0.398 (0.3024) | 0.207 (0.1744) | 0.144 (0.1254) | 0.236 (0.3163)

24. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: 12-lead ECG was measured in a semi-supine position using an automated ECG machine. Abnormal findings were categorized as clinically significant (CS) and not clinically significant (NCS). Data for any time till end of study were presented.
Time Frame: Up to 10 years and 11 months
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 16 | 6 | 12
Participants
  Abnormal, not clinically significant | 4 | 14 | 3 | 9
  Abnormal, clinically significant | 0 | 2 | 1 | 3

25. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Female: Follicle Stimulating Hormone (FSH) and Luteinizing Hormone (LH) at End of Study
Description: FSH and LH level of participants were measured. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 3 | 6 | 3 | 7
International units per Liter
  FSH | 0.200 (1.2490) | 3.217 (4.0455) | 0.100 (3.6042) | -0.336 (3.7053)
  LH | 0.03 (0.058) | 5.17 (9.665) | 4.17 (9.563) | 0.61 (9.778)

26. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Female: Follicle Stimulating Hormone (FSH) and Luteinizing Hormone (LH) at 20 Years of Age of Participants
Description: FSH and LH level of participants were measured. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529.Change from Baseline was calculated by subtracting the Baseline value from the specified time point value. Only participants with data at 20 year visit is presented. When participants reached pubertal maturity prior to being 20 years of age then these tests were not repeated at 20-years of age of participants.
Time Frame: Baseline (Day 1) and at 20 years of age of participants
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 1 | 3 | 1 | 3
International units per Liter
  FSH | 35.800 (NA) — NA indicates standard deviation could not be calculated due to single participant | 0.800 (1.2530) | -2.500 (NA) — NA indicates standard deviation could not be calculated due to single participant | 0.967 (0.3055)
  LH | 8.60 (NA) — NA indicates standard deviation could not be calculated due to single participant | 6.17 (16.717) | -6.30 (NA) — NA indicates standard deviation could not be calculated due to single participant | 5.10 (4.597)

27. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Female: Inhibin B at End of Study
Description: Inhibin B level of participants was measured. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed. At end of study, participants did not receive Ambrisentan 7.5 mg dose for evaluation of Inhibin B hence N=0
Measure: Mean (Standard Deviation); unit: Nanogram per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 2 | 5 | 0 | 4
Nanogram per liter | 0.0 (11.31) | 14.0 (67.48) |  | -29.0 (27.60)

28. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Female: Inhibin B at 20 Years of Age of Participants
Description: Inhibin B level of participants was measured. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529.Change from Baseline was calculated by subtracting the Baseline value from the specified time point value. Only participants with data at 20 year visit is presented. When participants reached pubertal maturity prior to being 20 years of age then these tests were not repeated at 20-years of age of participants.
Time Frame: Baseline (Day 1) and at 20 years of age of participants
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 1 | 2 | 1 | 2
Nanogram per liter | 0.0 (NA) — NA indicates standard deviation could not be calculated due to single participant | 49.0 (110.31) | 37.0 (NA) — NA indicates standard deviation could not be calculated due to single participant | 7.5 (70.00)

29. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Female: Sex Hormone Binding Globulin at End of Study
Description: Sex hormone binding globulin level of participants was measured. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 2 | 6 | 2 | 4
Nanomoles per liter | -10.0 (1.41) | 11.8 (14.22) | 0.5 (0.71) | 17.3 (22.31)

30. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Female: Sex Hormone Binding Globulin at 20 Years of Age of Participants
Description: Sex hormone binding globulin level of participants was measured. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Only participants with data at 20 year visit is presented. When participants reached pubertal maturity prior to being 20 years of age then these tests were not repeated at 20-years of age of participants.
Time Frame: Baseline (Day 1) and at 20 years of age of participants
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 1 | 3 | 1 | 2
Nanomoles per liter | 49.0 (NA) — NA indicates standard deviation could not be calculated due to single participant | 1.7 (54.37) | 10.0 (NA) — NA indicates standard deviation could not be calculated due to single participant | -15.5 (2.12)

31. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Female: Estrone at End of Study
Description: Estrone level of female participants was measured. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomole per milliliter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 1 | 5 | 2 | 5
Picomole per milliliter | 0.00 (NA) — NA indicates standard deviation could not be calculated due to single participant | -6.80 (178.361) | -26.00 (209.304) | 17.00 (125.913)

32. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Female: Estrone at 20 Years of Age of Participants
Description: Estrone level of female participants was measured. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529.Change from Baseline was calculated by subtracting the Baseline value from the specified time point value. Only participants with data at 20 year visit is presented. When participants reached pubertal maturity prior to being 20 years of age then these tests were not repeated at 20-years of age of participants.
Time Frame: Baseline (Day 1) and at 20 years of age of participants
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomole per milliliter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 1 | 2 | 1 | 2
Picomole per milliliter | -7.00 (NA) — NA indicates standard deviation could not be calculated due to single participant | 179.00 (196.576) | 11.00 (NA) — NA indicates standard deviation could not be calculated due to single participant | 89.00 (73.539)

33. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Female: Estriol at End of Study
Description: Estriol level of female participants will be measured. Only those parameters having status as overall will be presented. Baseline is the last value recorded prior to start of study treatment from AMB112529. Change from Baseline is calculated by subtracting the Baseline value from the end of study post-dose visit value. Data for this endpoint will be available for this endpoint by June 2023
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Reporting Status: Not Posted, anticipated posting 2023-06

34. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Female: Estriol at 20 Years of Age of Participants
Description: Estriol level of female participants will be measured. Only those parameters having status as overall will be presented. Baseline is the last value recorded prior to start of study treatment from AMB112529.Change from Baseline is calculated by subtracting the Baseline value from the specified time point value. Only participants with data at 20 year visit is presented. When participants reached pubertal maturity prior to being 20 years of age then these tests were not repeated at 20-years of age of participants. Data for this endpoint will be available for this endpoint by June 2023
Time Frame: Baseline (Day 1) and at 20 years of age of participants
Reporting Status: Not Posted, anticipated posting 2023-06

35. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Female: Estradiol at End of Study
Description: Estradiol level of female participants was measured. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomoles per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 1 | 4 | 2 | 5
Picomoles per liter | -11.00 (NA) — NA indicates standard deviation could not be calculated due to single participant | -77.25 (211.435) | -255.50 (427.800) | 44.80 (264.452)

36. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Female: Estradiol at 20 Years of Age of Participants
Description: Estradiol level of female participants was measured. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529.Change from Baseline was calculated by subtracting the Baseline value from the specified time point value. Only participants with data at 20 year visit is presented. When participants reached pubertal maturity prior to being 20 years of age then these tests were not repeated at 20-years of age of participants.
Time Frame: Baseline (Day 1) and at 20 years of age of participants
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomoles per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 1 | 1 | 1 | 2
Picomoles per liter | 55.50 (NA) — NA indicates standard deviation could not be calculated due to single participant | -107.00 (NA) — NA indicates standard deviation could not be calculated due to single participant | 15.00 (NA) — NA indicates standard deviation could not be calculated due to single participant | 387.50 (375.474)

37. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Male: FSH and LH at End of Study
Description: as for outcome 25
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 1 | 3 | 2 | 2
International units per Liter
  FSH | 6.000 (NA) — NA indicates standard deviation could not be calculated due to single participant | 0.267 (0.3215) | 3.250 (3.4648) | 0.850 (2.4749)
  LH | 3.20 (NA) — NA indicates standard deviation could not be calculated due to single participant | 1.70 (1.473) | 3.55 (2.333) | 3.55 (4.738)

38. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Male: FSH and LH at 20 Years of Age of Participants
Description: as for outcome 26
Time Frame: Baseline (Day 1) and at 20 years of age of participants
Population: Safety Population. Only those participants with available data at the specified time points were analyzed. No male participants received Ambrisentan 2.5mg dose at the time of attaining 20 years of age, hence N=0; No endocrinology laboratory tests were performed for 5 mg dose at the 20-year visit, hence N=0.
Measure: Mean (Standard Deviation); unit: International unit per Liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 0 | 0 | 2 | 1
International unit per Liter
  FSH |  |  | 2.350 (3.6062) | 0.500 (NA) — NA indicates standard deviation could not be calculated due to single participant
  LH |  |  | 2.90 (2.828) | 0.60 (NA) — NA indicates standard deviation could not be calculated due to single participant

39. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Male: Inhibin B at End of Study
Description: as for outcome 27
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed. No participants were analyzed for evaluation of Inhibin B in Ambrisentan 2.5 mg arm, hence N=0
Measure: Mean (Standard Deviation); unit: Nanogram per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 0 | 2 | 2 | 2
Nanogram per liter |  | 15.0 (5.66) | 8.5 (6.36) | 73.0 (175.36)

40. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Male: Inhibin B at 20 Years of Age of Participants
Description: as for outcome 28
Time Frame: Baseline (Day 1) and at 20 years of age of participants
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Nanogram per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 0 | 0 | 2 | 1
Nanogram per liter |  |  | 23.0 (21.21) | -47.0 (NA) — NA indicates standard deviation could not be calculated due to single participant

41. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Male: Sex Hormone Binding Globulin at End of Study
Description: as for outcome 29
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed. At end of study, no participants were analyzed for evaluation of Sex harmone binding globulin in 2.5 mg dose, hence N=0
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 0 | 2 | 2 | 2
Nanomoles per liter |  | -28.5 (28.99) | -11.5 (3.54) | -11.0 (39.60)

42. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Male: Sex Hormone Binding Globulin at 20 Years of Age of Participants
Description: Sex hormone binding globulin level of participants was measured. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529.Change from Baseline was calculated by subtracting the Baseline value from the specified time point value. Only participants with data at 20 year visit is presented. When participants reached pubertal maturity prior to being 20 years of age then these tests were not repeated at 20-years of age of participants.
Time Frame: Baseline (Day 1) and at 20 years of age of participants
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 0 | 0 | 2 | 1
Nanomoles per liter |  |  | -2.5 (12.02) | 12.0 (NA) — NA indicates standard deviation could not be calculated due to single participant

43. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Male: Total Testosterone at End of Study
Description: Total Testosterone level of participants was measured. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 1 | 3 | 2 | 2
Nanomoles per liter | 10.650 (NA) — NA indicates standard deviation could not be calculated due to single participant | 2.900 (7.1190) | 7.300 (1.6971) | 17.175 (0.1061)

44. Primary Outcome: Change From Baseline in Plasma Endocrine Parameters - Male: Total Testosterone at 20 Years of Age of Participants
Description: Total Testosterone level of participants was measured. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529.Change from Baseline was calculated by subtracting the Baseline value from the specified time point value. Only participants with data at 20 year visit is presented. When participants reached pubertal maturity prior to being 20 years of age then these tests were not repeated at 20-years of age of participants.
Time Frame: Baseline (Day 1) and at 20 years of age of participants
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Nanomoles per liter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 0 | 0 | 2 | 1
Nanomoles per liter |  |  | 4.000 (10.7480) | 6.600 (NA) — NA indicates standard deviation could not be calculated due to single participant

45. Primary Outcome: Change From Baseline of Pubertal Development in Male: Testicular Volume at End of Study
Description: Testicular volume was assessed by Prader's orchiodometer and the assessment was performed by a pediatric endocrinologist using the Tanner's criteria. Only those parameters having status - overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value. Data reported for left and right testicular volume.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed. No participants were analyzed for evaluation of testicular volume in 2.5 mg dose, hence N=0
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 0 | 2 | 2 | 2
Milliliter
  Right TV: number analyzed (Participants) | 0 | 1 | 2 | 2
  Right TV |  | 0.0 (NA) — NA indicates standard deviation could not be calculated due to single participant | 15.0 (7.07) | 11.5 (16.26)
  Left TV |  | 6.0 (8.49) | 16.5 (4.95) | 13.0 (14.14)

46. Primary Outcome: Change From Baseline of Pubertal Development in Male: Testicular Volume at 20 Years of Age of Participants
Description: Testicular volume was assessed by Prader's orchiodometer and the assessment was performed by a pediatric endocrinologist using the Tanner's criteria. Only those parameters having status as overall were presented. Baseline was the last value recorded prior to start of study treatment from AMB112529.Change from Baseline was calculated by subtracting the Baseline value from the specified time point value. Only participants with data at 20 year visit is presented. When participants reached pubertal maturity prior to being 20 years of age then these tests were not repeated at 20-years of age of participants. Data reported for left and right testicular volume.
Time Frame: Baseline (Day 1) and at 20 years of age of participants
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 0 | 1 | 2 | 1
Milliliter
  Right TV: number analyzed (Participants) | 0 | 0 | 2 | 1
  Right TV |  |  | 15.0 (7.07) | 8.0 (NA) — NA indicates standard deviation could not be calculated due to single participant
  Left TV |  | 17.0 (NA) — NA indicates standard deviation could not be calculated due to single participant | 16.5 (4.95) | 8.0 (NA) — NA indicates standard deviation could not be calculated due to single participant

47. Primary Outcome: Time to Change in Dose of Ambrisentan or Other Targeted PAH Therapeutic Agents (Prostanoids, Phosphodiesterase Type 5 [PDE-5] Inhibitors) Due to Tolerability Issues
Description: Time to change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, Phosphodiesterase type 5 [PDE-5] inhibitors) due to tolerability issues was defined as the time from randomization to the first occurrence of a dose change due to tolerability issues.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: Safety Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 1 | 2 | 1 | 3
Days | 393.0 (NA) — NA indicates standard deviation could not be calculated due to single participant | 468.5 (41.72) | 354.0 (NA) — NA indicates standard deviation could not be calculated due to single participant | 1448.7 (745.09)

48. Secondary Outcome: Number of Participants With All-cause Death
Description: Number of participants with all-cause death is presented.
Time Frame: Up to 10 years and 11 months
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
Number analyzed (Participants) | 4 | 16 | 6 | 12
Participants | 0 | 4 | 1 | 2

49. Secondary Outcome: Change From Baseline in the 6 Minutes Walking Distance (6MWD) Test
Description: Participant's 6 MWD data has been presented into three categories as overall, with oxygen use and without oxygen use. The 6-minute walk test measures the distance that a participant can walk in 6 minutes. All participants were given standardized instructions and the distance walked was measured. Baseline which is the last value recorded prior to start of study treatment in AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: ITT Population consisted of all participants who received at least 1 dose of study drug. Participants were considered as belonging to their treatment group at the start of study AMB114588. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Ambrisentan 2.5 mg (ITT) | Ambrisentan 5 mg (ITT) | Ambrisentan 7.5 mg (ITT) | Ambrisentan 10 mg (ITT)
Number analyzed (Participants) | 9 | 11 | 4 | 5
Meters
  Overall | 98.53 (115.355) | 56.74 (58.069) | 3.05 (94.659) | 34.24 (72.135)
  With oxygen use: number analyzed (Participants) | 2 | 0 | 0 | 0
  With oxygen use | -13.05 (96.944) |  |  |
  Without oxygen use: number analyzed (Participants) | 7 | 11 | 4 | 5
  Without oxygen use | 130.41 (104.115) | 56.74 (58.069) | 3.05 (94.659) | 34.24 (72.135)

50. Secondary Outcome: Time to the First Clinical Worsening of PAH
Description: Time to clinical worsening of PAH is defined as the time from randomization to first occurrence of death (all cause), placed on active list for lung transplant, and/or atrial septostomy, hospitalization due to PAH deterioration, addition of another targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to deterioration of clinical condition, change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to deterioration of clinical condition, PAH related deterioration identified by increase in WHO functional class, deterioration in exercise testing (i.e., 20% decrease in 6MWD on two consecutive tests -1 week apart, clinical signs or symptoms of right sided heart failure (i.e., new peripheral edema, increase in liver size, ascites, increase in jugular venous pressure, pericardial effusion, increased dyspnea).
Time Frame: Up to 10 years and 11 months
Population: ITT Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ambrisentan 2.5 mg (ITT) | Ambrisentan 5 mg (ITT) | Ambrisentan 7.5 mg (ITT) | Ambrisentan 10 mg (ITT)
Number analyzed (Participants) | 2 | 5 | 3 | 1
Days | 315.5 (2.12) | 896.2 (721.33) | 1122.0 (704.09) | 228.0 (NA) — NA indicates standard deviation could not be calculated due to single participant

51. Secondary Outcome: Time to the Addition of Another Targeted PAH Therapeutic Agent Due to Deterioration of Clinical Condition
Description: Time to addition of another targeted PAH therapeutics agents due to deterioration of clinical condition was defined as the time from randomization to the first occurrence of deterioration of clinical condition.
Time Frame: Up to 10 years and 11 months
Population: ITT Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ambrisentan 2.5 mg (ITT) | Ambrisentan 5 mg (ITT) | Ambrisentan 7.5 mg (ITT) | Ambrisentan 10 mg (ITT)
Number analyzed (Participants) | 1 | 2 | 1 | 2
Days | 510.0 (NA) — NA indicates standard deviation could not be calculated due to single participant | 697.5 (863.38) | 909.0 (NA) — NA indicates standard deviation could not be calculated due to single participant | 345.5 (109.60)

52. Secondary Outcome: Time to the Addition of Another Targeted PAH Therapeutic Agent Due to Lack of Beneficial Effect With Previous Therapy
Description: The time to addition of another targeted PAH therapeutic agents due to lack of beneficial effect with previous therapy was defined as the time from randomization to the first occurrence of lack of beneficial effect with previous therapy (not reaching set treatment goals).
Time Frame: Up to 10 years and 11 months
Population: ITT Population. Only those participants with available data at the specified time points were analyzed. Participants in higher dose group (7.5 and 10 mg) were not taking any additional therapeutic PAH agent hence N=0.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ambrisentan 2.5 mg (ITT) | Ambrisentan 5 mg (ITT) | Ambrisentan 7.5 mg (ITT) | Ambrisentan 10 mg (ITT)
Number analyzed (Participants) | 2 | 1 | 0 | 0
Days | 315.5 (2.12) | 173.0 (NA) — NA indicates standard deviation could not be calculated due to single participant |  |

53. Secondary Outcome: Time to Change in Dose of Ambrisentan or Other Targeted PAH Therapeutic Agents (Prostanoids, PDE-5 Inhibitors) Due to Deterioration of Clinical Condition
Description: Time to change in dose of ambrisentan or other targeted PAH therapeutic agents (prostanoids, PDE-5 inhibitors) due to deterioration of clinical condition was defined as the time from randomization to the first occurrence of a dose change due to deterioration of clinical condition.
Time Frame: Up to 10 years and 11 months
Population: ITT Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ambrisentan 2.5 mg (ITT) | Ambrisentan 5 mg (ITT) | Ambrisentan 7.5 mg (ITT) | Ambrisentan 10 mg (ITT)
Number analyzed (Participants) | 3 | 3 | 1 | 2
Days | 1247.3 (1051.97) | 1097.0 (922.77) | 909.0 (NA) — NA indicates standard deviation could not be calculated due to single participant | 345.5 (109.60)

54. Secondary Outcome: Change From Baseline in Subject Global Assessment (SF-10) Health Survey for Children
Description: The short-form 10 (SF-10) Health Survey for children is a 10-item, 4-week recall, parent-completed health assessment that measures physical and psychosocial functioning for children ages five and over. Two summary scores were calculated: a Physical Summary Score (PHS) and a Psychosocial Summary Score (PSS) with a range of 5 to 30 points for each 5-item score. The aggregate score was then standardized and transformed to a norm-based scoring metric in accordance with the developer's guidelines. This generated the final standardized norm-based scores for PHS (range -10.90 to 57.21) and for PSS (range 8.81 to 62.28), respectively. A higher value on each summary score indicates better functioning. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: ITT Population. Only those participants with available data at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ambrisentan 2.5 mg (ITT) | Ambrisentan 5 mg (ITT) | Ambrisentan 7.5 mg (ITT) | Ambrisentan 10 mg (ITT)
Number analyzed (Participants) | 8 | 9 | 4 | 5
Scores on a scale
  Physical health summary | -1.618 (7.4650) | -0.967 (16.4890) | -1.788 (12.0104) | -0.272 (15.1029)
  Psychosocial summary | -0.336 (5.4290) | -1.880 (7.9810) | 2.225 (6.2357) | 6.766 (6.5080)

55. Secondary Outcome: Number of Participants With Change From Baseline in World Health Organization (WHO) Functional Class of PAH
Description: PAH was classified by WHO functional class (FC) at specific time points. There were four WHO FC grades based on severity of PAH symptoms (Class I=none, Class IV=most severe). Grades were mapped to numeric scale for which scores ranged from 1-4 (i.e. Class I=1 and IV=4). Change categorization was based on change from Baseline scores: -2, -1, 0, +1, +2. Data was categorized as No Change (0), Improved (-1,-2), Deteriorated (+1,+2). Baseline was the last value recorded prior to start of study treatment from AMB112529. Higher score indicated higher severity.Change from Baseline was calculated by subtracting the Baseline value from the end of study post-dose visit value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: ITT Population. Only those participants with available data at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ambrisentan 2.5 mg (ITT) | Ambrisentan 5 mg (ITT) | Ambrisentan 7.5 mg (ITT) | Ambrisentan 10 mg (ITT)
Number analyzed (Participants) | 9 | 11 | 4 | 5
Participants
  Improved | 5 | 5 | 3 | 0
  No Change | 4 | 6 | 1 | 5
  Deteriorated | 0 | 0 | 0 | 0

56. Secondary Outcome: Percentage Change From Baseline in Plasma N-terminal Pro-B-type Natriuretic Peptide (NT-Pro BNP) Concentration
Description: Blood samples were collected to analyze NT-Pro BNP concentration at specific time points. Baseline was the last value recorded prior to start of study treatment from AMB112529. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline (Day 1) and up to 10 years and 11 months
Population: ITT Population. Only those participants with available data at the specified time points were analyzed.
Measure: Geometric Mean (Full Range); unit: Percentage Change
Arm/Group | Ambrisentan 2.5 mg (ITT) | Ambrisentan 5 mg (ITT) | Ambrisentan 7.5 mg (ITT) | Ambrisentan 10 mg (ITT)
Number analyzed (Participants) | 7 | 11 | 2 | 5
Percentage Change | -62.59 [-97.6 to 116.3] | -56.02 [-99.0 to 2227.1] | 59.06 [-22.6 to 226.8] | 101.96 [-2.1 to 214.4]

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-STEAEs and STEAEs were collected from the start of study treatment up to 10 years and 11 months
Description: All-cause mortality, non-STEAEs and STEAEs were collected in Safety Population which consisted of all participants who received at least 1 dose of study drug. Participants were considered as belonging to the treatment group according to the highest dose received in the extension study (AMB114588).
Arm/Group | Ambrisentan 2.5 mg (Safety) | Ambrisentan 5 mg (Safety) | Ambrisentan 7.5 mg (Safety) | Ambrisentan 10 mg (Safety)
All-Cause Mortality (participants affected / at risk) | 0/4 | 4/16 | 1/6 | 2/12
Serious Adverse Events (participants affected / at risk) | 2/4 | 7/16 | 4/6 | 8/12
Other Adverse Events (participants affected / at risk) | 3/4 | 13/16 | 5/6 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambrisentan 2.5 mg (Safety) (N=4) | Ambrisentan 5 mg (Safety) (N=16) | Ambrisentan 7.5 mg (Safety) (N=6) | Ambrisentan 10 mg (Safety) (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wandering pacemaker (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Autoimmune lymphoproliferative syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambrisentan 2.5 mg (Safety) (N=4) | Ambrisentan 5 mg (Safety) (N=16) | Ambrisentan 7.5 mg (Safety) (N=6) | Ambrisentan 10 mg (Safety) (N=12)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conductive deafness (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Astigmatism (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (5) | 2 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site discharge (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Puncture site pain (General disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 2 (3) | 2 (2)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to vaccine (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Immunisation reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (7) | 1 (1) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 2 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 5 (18) | 1 (3) | 3 (9)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (3)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pharyngitis (Infections and infestations) | 1 (2) | 3 (4) | 0 (0) | 2 (4)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 1 (4)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (4) | 3 (8) | 4 (7) | 2 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood parathyroid hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 2 (3) | 2 (7)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tardive dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device leakage (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Automatism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erection increased (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Therapeutic procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cyanosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT01342952/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT01342952/SAP_001.pdf